CLINICAL TRIAL: NCT04830410
Title: The Effects of Fructans in Irritable Bowel Syndrome
Brief Title: The Effects of Carbohydrates in Irritable Bowel Syndrome
Acronym: FIBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Atmo Biosciences Pty Ltd (Industry); Beneo-Institute (Industry)
Responsible Party: Principal Investigator, Magnus Simrén, Professor, Göteborg University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FIBS 2020-03644
Record Dates: First submitted 2021-03-26; First posted 2021-04-05 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
Keywords: Fructans; FODMAP; carbohydrates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: After a low FODMAP diet, patients will have to reintroduce fructan or placebo powder. Patients will be randomized by a web-mail randomization.The powder bags were prepared and named A or B by the firms Beneo, and the participants and the staff involved in the study will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fructan powder (Experimental): 2 g of fructan powder 3 times per day for 7 days
  Interventions: Dietary Supplement: Fructan reintroduction
- Placebo (Placebo Comparator): 2g of placebo (maltodextrin) 3 times per day for 7 days.
  Interventions: Dietary Supplement: Placebo reintroduction

INTERVENTIONS:
Dietary Supplement: Fructan reintroduction — Patients will reintroduce fructan powder after 14-day of a low FODMAP diet
  Arms: Fructan powder
Dietary Supplement: Placebo reintroduction — Patients will reintroduce placebo powder after 14-day of a low FODMAP diet
  Arms: Placebo

SUMMARY:
Food and their components are often reported as gastrointestinal (GI) symptom triggers in patients with IBS. The current interest in dietary management in IBS, has largely focused on the negative effect of poorly absorbed and subsequently fermented carbohydrates (FODMAP - Fermentable Oligo-, Di-, Mono-saccharides And Polyols). These unabsorbed carbohydrates can generate GI symptoms through osmosis, with increased amount of fluid in the gut lumen, and via modification of gut microbiota composition and function (fermentation and production of gas).

Studies assessing diets low in FODMAPs have shown promising results in symptom improvement in some IBS patients, but not in all. The low FODMAP diet, as it is used today, is restrictive and difficult for patients to accommodate in their daily life. Moreover, the effect of this diet on microbiota composition and function is not defined, and there are also concerns that restrictive diets may lead to nutritional inadequacy.

Fructan is a specific FODMAP which is built of fructose polymers. Examples of foods that contain fructans are wheat, onion, garlic and banana. The daily dietary intake of fructans varies approximately between 3 and 6 grams. Fructans are potential triggers of GI symptoms in IBS however, they are currently also used as prebiotic supplements. A recent systematic review and meta-analysis concluded that low dosages of fructans do not worsen GI symptoms, but they do increase the beneficial bifidobacteria. It remains unclear whether the potential benefits of fructans outweigh the potential harmful effects in patients with IBS.

The investigators are aiming to assess the effects of fructans, as well as predictive factors and mechanisms involved, and to compare with placebo in IBS patients. The investigators will assess GI symptom severity, visceral sensitivity, intestinal gas production, gut immunity and microbiota, and metabolites produced in the gut.

ELIGIBILITY:
Inclusion Criteria:

* IBS according to ROME IV criteria (with diarrhoea)

Exclusion Criteria:

* Celiac disease or any other gastroenterology disease (such as inflammatory bowel disease, celiac disease, microscopic colitis, diverticulitis, radiation enteritis).
* Suspected or known strictures, fistulas or physiological/mechanical GI obstruction, history of gastric bezoar.
* Appendicectomy and cholecystectomy <3 months.
* Heart-, liver-, neurological-, or current psychiatric disease, diabetes, obesity (BMI>30), other disease or surgery to the abdomen that affected intestinal function.
* Implantable or portable electro-mechanical medical devices, e.g. pacemakers.
* Swallowing disorders/dysphagia to food or pills.
* Allergy or intolerances to foods.
* Compliance to a special diet (including vegan, vegetarian, gluten-free or low FODMAP diet).
* Pregnant or breast feeding.
* Usage of antibiotics within 4 weeks prior to inclusion
* Usage of alcohol more than 14 units per week.
* No new pharmacological treatment during the study period.
* Medications: laxatives, neuromodulators or opioids (morphine, codeine, tramadol…)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
IBS-SSS | before and after the reintroduction (7days +/-3 days)
  change in irritable bowel syndrome severity scoring system (IBS-SSS) between the 2 groups. IBS-SSS is between 0 and 500, with a higher score meaning more severe symptoms.

SECONDARY OUTCOMES:
visceral sensitivity | Baseline
  measured by a rectal barostat, predictor for a better GI response to a low FODMAP diet and predictor of a worse GI response to fructan reintroduction
change in intestinal gas production | between baseline and after (7days +/-3 days) of reintroduction
  measured by a gas sensing capsule (Atmo), between the 2 groups
change in gas production | between baseline and after (7days +/-3 days) of reintroduction
  measured by breath tests (H2 and CH4) between the 2 groups.
change in microbiota | between baseline, after the low FODMAP diet (14 days) and after reintroduction (7+/-3 days)
  Fecal microbiota analysis using 16S technique between the 2 groups.
Change in metabolomics profiles | between baseline, after the low FODMAP diet (14 days) and after reintroduction (7+/-3 days)
  Targeted and untargeted metabolomics in urine, blood and stool samples measured by Liquid and gas chromatography-mass spectrometry between the 2 groups.
change in stool form and frequency | between baseline, after the low FODMAP diet (14 days) and after reintroduction (7+/-3 days)
  Stool diary between the 2 groups.
GSRS-IBS | between baseline, after the low FODMAP diet (14 days) and after reintroduction (7+/-3 days)
  change in Gastrointestinal symptom rating scale-IBS (GSRS-IBS) between the 2 groups. GSRS-IBS assesses five GI symptom domains: satiety, abdominal pain, diarrhea, constipation and bloating. The five domains are calculated using the mean of two to four items scored with 7-point Likert scales, with higher scores representing more severe symptoms.
HAD | between baseline, after the low FODMAP diet (14 days) and after reintroduction (7+/-3 days)
  change in Hospital Anxiety and depression scale (HAD) between the 2 groups. HAD assesses the severity of psychological distress, i.e. anxiety and depression. In this 14-item scale, seven items measure anxiety and the other seven measure depression on a 4-point Likert scale (0-3) which provides a score between 0 (absence) and 21 (high level). Scores higher than 10 on each of the subscales is considered to define clinically relevant anxiety and/or depression.
VSI | between baseline, after the low FODMAP diet (14 days) and after reintroduction (7+/-3 days)
  change in Visceral sensitivity index (VSI) between the 2 groups. VSI is a 15-item validated scale measuring GI symptom-specific anxiety, i.e. the cognitive, affective, and behavioural response to fear of GI sensations, symptoms, and the context in which these occur. The total score ranges between 0 (no GI-specific anxiety) to 75 (severe GI-specific anxiety).
IBSQOL | between baseline, after the low FODMAP diet (14 days) and after reintroduction (7+/-3 days)
  change in irritable bowel syndrome quality of life (IBSQOL) questionnaire between the 2 groups. IBSQOL is a disease-specific, self-administered questionnaire, with 30 items measuring nine aspects of health-related quality of life during the past four weeks. The nine domains are emotional health, mental health, sleep, energy, physical functioning, food/diet, social role, physical role and sexual relations. Each question has five or six response options. For each subscale, the score is transformed to a 0-100 scale. A higher score represents a better quality of life.
PHQ12 | between baseline, after the low FODMAP diet (14 days) and after reintroduction (7+/-3 days)
  change in patient health questionnaire 12 (PHQ12) between the 2 groups. The PHQ-15 is a somatic symptom subscale derived from the full PHQ. It inquires about 15 somatic symptoms; each individual symptom is coded as 0, 1, or 2, and the total score ranges from 0 to 30, with higher scores representing more severe symptoms.
CSI | between baseline, after the low FODMAP diet (14 days) and after reintroduction (7+/-3 days)
  change in Central Sensitization Inventory (CSI) between the 2 groups. The responses were graded on a Likert scale from 0 (never) to 4 (always). The total score ranges from 0 to 100. A higher score suggest higher central sensitization syndrome.
IBS-SSS | between baseline, after the low FODMAP diet (14 days) and after reintroduction (7+/-3 days)
  change in irritable bowel syndrome severity scoring system (IBS-SSS) between the 2 groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided